CLINICAL TRIAL: NCT01433640
Title: Evaluation of Contrast-enhanced Mammography and Contrast-enhanced Breast Tomosynthesis: Comparison to Contrast-enhanced Breast MRI- A Pilot Study
Brief Title: Dual-energy Contrast-enhanced (2D and 3D Mammography Versus Contrast-enhanced MRI)- A Pilot Study
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-01
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: image on multi-modalities; visualize cancer lesions; highly suspicious lesions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Contrast-enhanced Mammography: Subjects will undergo 2D imaging with iodine contrast.
- Contrast-enhanced Breast Tomosynthesis: Subjects will undergo 3D imaging with iodine contrast.
- Contrast-enhanced MRI: Each subject imaged with iodine contrast will also be imaged with contrast-enhanced MRI using gadolinium.

SUMMARY:
This is a pilot study to evaluate 2D contrast-enhanced mammography image and 3D (tomosynthesis) contrast-enhanced images to contrast enhanced MRI in women with greater than 95% probability of breast cancer (BIRADS 5) or confirmed breast cancer (BIRADS 6).This study will then be used to design additional studies.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female of any race and ethnicity.
* Subject is at least 25 years old
* Subject has or will have a contrast enhanced breast MRI +/- 31 days of enrollment with no interval treatment or procedure between the two studies
* Subject has BIRADS 6 or BIRADS 5 cancer or as determined by the radiologist
* >50% of the biopsied cancer mass must remain following biopsy OR
* A calcification must be at least 2cm in maximum dimension prior to biopsy or at least 1cm in maximum dimension following biopsy

Exclusion Criteria:

* Subject is unable or unwilling to undergo informed consent
* Subject has breast implant in the breast to be imaged
* Subject is pregnant
* Subject is breast feeding or lactating
* Subject has a known allergy to gadolinium contrast agents.
* Subject has a contraindication for MRI.
* Subject suspected to be at risk to complication from the contrast agents.
* Subject has a documented renal insufficiency,
* Subject requires renal dialysis.
* Subject has had a prior reaction to iodinated contrast.
* Subject has had a prior episode of anaphylactic reaction to any substance.
* Subject has taken metformin (Glucophage) within 48 hours of study procedures.
* Subject has multiple allergies and/or severe asthma regularly treated with medication (prescription and/or over-the-counter).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes females of any race and ethnicity. The subjects must ba at least 25 years old and has a lesion of BIRADS 5 or BIRADS 6 as determined by a radiologist.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
A PILOT study to determine Cancer lesion enhancement with CEM and CEBT is non-inferior to that of CEMRI. | Fall 2012
  This Pilot study is designed to evaluate two x-ray contrast methods with contrast enhanced MRI. Each subject will be imaged with CEM, CEBT and CEMRI. The goals for this will be to:
  i) Using a Likert scale, Compare the enhancement of breast cancer lesions with CEM, CEBT and CEMRI.
  ii) Using a Likert scale, Compare the enhancement of benign breast lesions with CEM, CEBT and CEMRI.
  The results of this study will be used to design studies to measure the sensitivity and specificity of CEM and CEBT.

SECONDARY OUTCOMES:
Comparison of lesion conspicuity | up to one year post study enrollment
  Using a Likert scale the CEM and the CBT images will be compared with standard pre-contrast mammography and tomosynthesis images to determine lesion conspicuity.

CONTACTS AND LOCATIONS:
Overall Officials: John Lewins, MD, Principal Investigator — Rose Breast Center
Locations (1):
- Rose Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Weidner N, Semple JP, Welch WR, Folkman J. Tumor angiogenesis and metastasis--correlation in invasive breast carcinoma. N Engl J Med. 1991 Jan 3;324(1):1-8. doi: 10.1056/NEJM199101033240101. PMID 1701519
- [Background] Weidner N. The importance of tumor angiogenesis: the evidence continues to grow. Am J Clin Pathol. 2004 Nov;122(5):675-7. doi: 10.1309/KY6E-H0LG-Y6D6-PGP5. No abstract available. PMID 15491962
- [Background] Lehman CD, Gatsonis C, Kuhl CK, Hendrick RE, Pisano ED, Hanna L, Peacock S, Smazal SF, Maki DD, Julian TB, DePeri ER, Bluemke DA, Schnall MD; ACRIN Trial 6667 Investigators Group. MRI evaluation of the contralateral breast in women with recently diagnosed breast cancer. N Engl J Med. 2007 Mar 29;356(13):1295-303. doi: 10.1056/NEJMoa065447. Epub 2007 Mar 28. PMID 17392300
- [Background] Lindfors KK, Boone JM, Nelson TR, Yang K, Kwan AL, Miller DF. Dedicated breast CT: initial clinical experience. Radiology. 2008 Mar;246(3):725-33. doi: 10.1148/radiol.2463070410. Epub 2008 Jan 14. PMID 18195383
- [Background] Chen SC, Carton AK, Albert M, Conant EF, Schnall MD, Maidment AD. Initial clinical experience with contrast-enhanced digital breast tomosynthesis. Acad Radiol. 2007 Feb;14(2):229-38. doi: 10.1016/j.acra.2006.10.022. PMID 17236995
- [Background] Carton AK, Gavenonis SC, Currivan JA, Conant EF, Schnall MD, Maidment AD. Dual-energy contrast-enhanced digital breast tomosynthesis--a feasibility study. Br J Radiol. 2010 Apr;83(988):344-50. doi: 10.1259/bjr/80279516. Epub 2009 Jun 8. PMID 19505964
- [Background] Lewin JM, Isaacs PK, Vance V, Larke FJ. Dual-energy contrast-enhanced digital subtraction mammography: feasibility. Radiology. 2003 Oct;229(1):261-8. doi: 10.1148/radiol.2291021276. Epub 2003 Jul 29. PMID 12888621
- [Background] Jong RA, Yaffe MJ, Skarpathiotakis M, Shumak RS, Danjoux NM, Gunesekara A, Plewes DB. Contrast-enhanced digital mammography: initial clinical experience. Radiology. 2003 Sep;228(3):842-50. doi: 10.1148/radiol.2283020961. Epub 2003 Jul 24. PMID 12881585
- [Background] Diekmann F, Diekmann S, Jeunehomme F, Muller S, Hamm B, Bick U. Digital mammography using iodine-based contrast media: initial clinical experience with dynamic contrast medium enhancement. Invest Radiol. 2005 Jul;40(7):397-404. doi: 10.1097/01.rli.0000167421.83203.4e. PMID 15973130